CLINICAL TRIAL: NCT03382574
Title: Pilot Study of Denosumab in BRCA1/2 Mutation Carriers Scheduled for Risk-Reducing Salpingo-Oophorectomy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: it was decided that due to lack of accrual on the trial, and low potential for accruing over the near future, the trial will be shut down.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-02314; NCI-2017-02314 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAAR6281; N01-CN-2012-00034; AAAR6281 (Other: M D Anderson Cancer Center); MDA2017-09-03 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH); 2018-0478 (Other: MD Anderson Cancer Center ID)
Record Dates: First submitted 2017-12-22; First posted 2017-12-26 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Denosumab; QL1206; Salpingo-oophorectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (denosumab, risk-reducing salpingo-oophorectomy) (Experimental): Beginning within 3 days of menstrual cycle, patients receive denosumab SC every 4 weeks for 1-2 doses and undergo risk-reducing salpingo-oophorectomy 14-28 days after last dose.
  Interventions: Biological: Denosumab; Procedure: Salpingo-Oophorectomy
- Arm II (risk-reducing salpingo-oophorectomy) (Active Comparator): Patients receive no treatment for 2-8 weeks and then undergo risk-reducing salpingo-oophorectomy.
  Interventions: Procedure: Salpingo-Oophorectomy

INTERVENTIONS:
Biological: Denosumab — Given SC
  Other Names: AMG 162; AMG-162; Denosumab Biosimilar MW032; Denosumab Biosimilar QL1206; Denosumab Biosimilar TK-006; Prolia; TK-006; Xgeva
  Arms: Arm I (denosumab, risk-reducing salpingo-oophorectomy)
Procedure: Salpingo-Oophorectomy — Undergo risk-reducing salpingo-oophorectomy

SUMMARY:
This randomized pilot early phase I trial studies how well denosumab works in BRCA1/2 mutations carriers scheduled for risk-reducing salpingo-oophorectomy. Denosumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the effect of denosumab 120 mg subcutaneously every 4 weeks for 1-2 doses to no treatment in the pre-surgical setting on Ki67 proliferation index by immunohistochemistry (IHC) in the fimbrial end of the fallopian tube of premenopausal BRCA1/2 mutation carriers undergoing risk-reducing salpingo-oophorectomy, with or without hysterectomy.

SECONDARY OBJECTIVES:

I. To assess Ki67 proliferation index by immunohistochemistry (IHC) in ovarian surface epithelium and endometrium (if also undergoing a hysterectomy, ~20% of participants) after exposure to denosumab compared to no treatment.

II. To investigate other tissue-based biomarkers in the fimbrial end of the fallopian tube, ovarian surface epithelium, and endometrium (if also undergoing hysterectomy) after exposure to denosumab compared to no treatment, including:

IIa. Apoptosis with cleaved caspase-3 by IHC. IIb. Receptor activator of NF-KB (RANK) and RANK ligand (RANKL) expression by IHC.

IIc. Estrogen receptor (ER) and progesterone receptor (PR) expression by IHC. IId. CD44 and p53 expression by IHC. IIe. Signal transducer and activator of transcription 3 (STAT3) and phosphorylated-STAT3 (pSTAT3) expression by IHC.

III. To analyze gene expression profiling in the fimbrial end of the fallopian tube and ovarian surface epithelium after exposure to denosumab compared to no treatment.

IV. To investigate serum biomarkers at baseline (pre-treatment) and time of surgery (post-treatment) with denosumab compared to no treatment, including:

IVa. Progesterone. IVb. Estradiol. IVc. Denosumab drug levels. V. To investigate serial serum C-terminal telopeptide (CTX) levels from baseline (pre-treatment) to time of surgery to 9 months and 12 months after start of intervention with denosumab compared to no treatment.

VI. To monitor safety and adverse effects of denosumab compared to no treatment.

OUTLINE: Patients are randomized 1 of 2 arms.

ARM I: Beginning within 3 days of menstrual cycle, patients receive denosumab subcutaneously (SC) every 4 weeks for 1-2 doses and undergo risk-reducing salpingo-oophorectomy 14-28 days after last dose.

ARM II: Patients receive no treatment for 2-8 weeks and then undergo risk-reducing salpingo-oophorectomy.

After completion of study treatment, patients are followed up at 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be premenopausal (defined as < 3 months since last menstrual period OR serum follicle-stimulating hormone [FSH] < 20 mIU/mL)
* Documented germline pathogenic or likely pathogenic variant in the BRCA1 or BRCA2 genes
* Participants must be scheduled for or in the process of scheduling a risk-reducing salpingo-oophorectomy with or without hysterectomy - either bilateral or unilateral (if prior unilateral oophorectomy or salpingectomy for benign condition)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT])) =< 1.5 x institutional ULN
* Creatinine clearance >= 30 mL/min
* Serum calcium or albumin adjusted >= 8.0 mg/dL and =< 11.5 mg/dL
* Participant must have a negative urine or serum pregnancy test 14 days prior to randomization or drug administration; the effects of denosumab on the developing human fetus at the recommended therapeutic dose may cause fetal harm when administered to pregnant women; women of childbearing potential must agree to use adequate contraception from time of drug administration to time of surgery; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Women currently on hormonal contraception (i.e., oral contraceptives, Mirena intrauterine device [IUD]) are eligible to participate if they have been on a stable dose for at least 3 months; women who have undergone bilateral tubal ligation are also eligible to participate in this study; there will be stratification for hormonal contraceptive use within 3 months prior to registration
* Participants must be willing to take supplemental oral calcium 1000 mg (two 500 mg tablets) and vitamin D3 1000 IU daily for six months (which will be supplied by the research study) after receiving denosumab treatment or no treatment
* Ability to understand and the willingness to sign a written informed consent document in English or Spanish or Hebrew
* Participants must have a dental examination =< 6 months of study registration
* Willing to not undergo any other elective surgery procedure with general anesthesia or conscious sedation during the treatment period; the treatment period is completed after the last injection of denosumab is administered

Exclusion Criteria:

* History of ovarian cancer; history of breast cancer or any other malignancy is permitted if last chemotherapy treatment was greater than 6 months prior to registration and participant is not using endocrine therapy
* Previous treatment with denosumab (including Prolia for osteoporosis or Xgeva for bone metastases) or use of bisphosphonate within 3 months of registration to the study
* Participants receiving any other investigational agents
* History of allergic reactions or hypersensitivity attributed to denosumab or any components of denosumab or compounds of similar chemical or biologic composition to denosumab, such as other RANKL inhibitors
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study because denosumab is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with denosumab, breastfeeding should be discontinued if the mother is treated with denosumab; there is no minimum amount of time since pregnancy/breastfeeding required before enrolling into the study; however, the date of delivery, pregnancy termination, or weaning from breastfeeding will be documented on case report forms; female subjects of child bearing potential and not willing to use, in combination with her partner, highly effective contraception during treatment will be excluded
* Use of endocrine therapy (selective estrogen receptor modulator, aromatase inhibitor, gonadotrophin releasing hormone [GnRH] agonist) within 6 months of registration to the study
* Prior history or current evidence of osteonecrosis or osteomyelitis of the jaw, evidence of untreated local gum or oral infection, or non-healed dental or oral surgery
* Active dental or jaw conditions which require oral surgery/dental procedures, including tooth extraction within 6 months of registration to the study; dental fillings are permitted within 6 months of study registration
* Other risk factors for the development of osteonecrosis of the jaw (ONJ) including poor oral hygiene, use of a dental appliance, immunosuppressive therapy, treatment with angiogenesis inhibitors, systemic corticosteroids, diabetes, or gingival infections
* Known sensitivity to any of the products to be administered during the study (e.g., calcium or vitamin D)
* Known serious infections, including a history of active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV); screening for these infections is not required for study enrollment
* Hypocalcemia (serum calcium or albumin adjusted calcium < 8.0 mg/dL) or renal dysfunction (creatinine clearance < 30 mL/min)
* Women with known osteoporosis or history of osteoporotic (fragility) fracture of the spine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Powel Brown, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas
- Israel (2):
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter protocol will be conducted at the following five sites: Columbia University Irving Medical Center (CUIMC), New York, NY; Weill-Cornell Medical Center, New York, NY; the Dana Farber Cancer Institute (DFCI), Boston, MA; and Tel Aviv Sourasky Medical Center and Chaim Sheba Medical Center, Tel Aviv, Israel.
Pre-assignment Details: 2 participants consented at Tel Aviv Sourasky Medical Center, no participants randomized nor received trial intervention (Participant 1 was deemed ineligible due to elevated FSH level and Participant 2 did not start intervention due to COVID-19 lockdown restrictions).
Groups:
- Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy)/Arm II (Risk-reducing Salpingo-oophorectomy): Beginning within 3 days of menstrual cycle, patients receive denosumab SC every 4 weeks for 1-2 doses and undergo risk-reducing salpingo-oophorectomy 14-28 days after last dose.
  Denosumab: Given SC
  Salpingo-Oophorectomy: Undergo risk-reducing salpingo-oophorectomy
  Arm II Patients receive no treatment for 2-8 weeks and then undergo risk-reducing salpingo-oophorectomy.
  Salpingo-Oophorectomy: Undergo risk-reducing salpingo-oophorectomy
Period: Overall Study
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy)/Arm II (Risk-reducing Salpingo-oophorectomy)
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 2 participants consented at Tel Aviv Sourasky Medical Center, no participants randomized nor received trial intervention combined arms due to the participants were not randomized.
Groups:
- Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy)/ Arm II (Risk-reducing Salpingo-oophorectomy): Beginning within 3 days of menstrual cycle, patients receive denosumab SC every 4 weeks for 1-2 doses and undergo risk-reducing salpingo-oophorectomy 14-28 days after last dose.
  Denosumab: Given SC
  Salpingo-Oophorectomy: Undergo risk-reducing salpingo-oophorectomy
  Arm II Patients receive no treatment for 2-8 weeks and then undergo risk-reducing salpingo-oophorectomy.
  Salpingo-Oophorectomy: Undergo risk-reducing salpingo-oophorectomy
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy)/ Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Ki67 Proliferation Index Fallopian Tube Fimbrial Epithelial Cells
Description: Will be assessed using immunohistochemistry (IHC). Quantitative measures of the expression of Ki67 based upon percentage of positive cells will be scored by a pathologist blinded to treatment assignment. In order to evaluate the difference of Ki67 expression between the two arms, 2-sample t-test will be considered.
Time Frame: Up to 12 months
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Ki67 Proliferation Index in Ovarian Surface Epithelium and Endometrium
Description: Will be assessed using IHC. In order to evaluate the difference of Ki67 expression between the two arms, 2-sample t-test will be considered.
Time Frame: Up to 12 months
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Other Tissue-based Biomarkers in the Fimbrial End of the Fallopian Tube, Ovarian Surface Epithelium, and Endometrium
Description: Will be assessed using IHC. Including: apoptosis with cleaved caspase-3 (IHC), RANK/RANKL (IHC), estrogen receptor (ER)/progesterone receptor (PR) (IHC), CD44 and p53 (IHC), and STAT3 and pSTAT3 (IHC). Values of tissue-based biomarkers measurements such as tissue Ki67 proliferation index, serum progesterone, etc., which are continuous variables, will be summarized by descriptive statistics including mean, standard deviation, median and range. For tissue biomarkers, linear regression models will be employed to investigate the association of treatment while adjusting for possible confounders (i.e., age, race, etc.). Normality, homoscedasticity, independence of errors, and lack of multicollinearity in the covariates will be evaluated; if needed, proper transformation will be considered.
Time Frame: Up to 12 months
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Gene Expression Profiling of RANK, Cell Proliferation, Cell Cycle Progression, and Inflammation Pathways
Description: For gene expression profiling analysis, nSolver Analysis Software (nanoString Technologies, Washington [WA]) will be used. Geometric mean is used for calculation of normalization factors. Student's t test is used to calculate differential expression.
Time Frame: Up to 12 months
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serum Biomarkers Including Progesterone, Estradiol, and Denosumab Drug Levels
Description: Values of serum biomarkers measurements such as tissue Ki67 proliferation index, serum progesterone, etc., which are continuous variables, will be summarized by descriptive statistics including mean, standard deviation, median and range.
Time Frame: Up to time of surgery
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Serial Serum C-terminal Telopeptide Levels
Description: 2-sample t-test may be applied to evaluate any change in serum biomarkers from baseline to after intervention. To investigate the overall changes in serum biomarkers, a linear mixed model that accommodates intra-participant correlation due to repeated measurements will be utilized adjusting for any potential covariates.
Time Frame: Baseline up to 12 months after start of intervention
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Toxicity Profile and Frequency of Adverse Effects in Premenopausal BRCA1/2 Mutation Carriers
Description: Categorical variables, such as adverse events, will be summarized by frequency and proportion.
Time Frame: Up to 12 months after start of treatment
Population: No participants were randomized, therefore no data collected.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: at baseline
Description: There were no adverse events because neither consented participant were randomized, so they never received trial intervention.
Arm/Group | Arm I (Denosumab, Risk-reducing Salpingo-oophorectomy) | Arm II (Risk-reducing Salpingo-oophorectomy)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03382574/Prot_SAP_000.pdf